CLINICAL TRIAL: NCT02824874
Title: A Randomized, Open-label, Multiple Dosing, 2-way Crossover Study to Evaluate the Effect of Sitagliptin on Pharmacokinetics of Lobeglitazone in Healthy Male Volunteers
Brief Title: CKD-396 Drug-drug Interaction Study(A) (CKD-396 DDI(A) P1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 165DDI16002
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1(Treatment A/Treatment B) (Experimental): Period 1: Treatment A(Duvie Tab. 0.5mg)*1T/day for 5 days, QD, PO
  Period 2: Treatment B(Duvie Tab. 0.5mg + Januvia Tab. 100mg)*1T/day for 5 dyas, QD, PO
  Each treatment period was separated by a washout period of at least 10 dyas.
  Interventions: Drug: Duvie Tab. 0.5mg; Drug: Duvie Tab. 0.5mg + Januvia Tab. 100mg
- Group 2(Treatment B/Treatment A) (Experimental): Period 1: Treatment B(Duvie Tab. 0.5mg + Januvia Tab. 100mg)*1T/day for 5 dyas, QD, PO
  Period 2: Treatment A(Duvie Tab. 0.5mg)*1T/day for 5 days, QD, PO
  Each treatment period was separated by a washout period of at least 10 dyas.
  Interventions: Drug: Duvie Tab. 0.5mg; Drug: Duvie Tab. 0.5mg + Januvia Tab. 100mg

INTERVENTIONS:
Drug: Duvie Tab. 0.5mg — Duvie Tab. 0.5mg*1T/day for 5days, QD, PO
  Other Names: Lobeglitazone 0.5mg
Drug: Duvie Tab. 0.5mg + Januvia Tab. 100mg — Duvie Tab. 0.5mg + Januvia Tab.100mg*1T/day for 5 dyas, QD, PO
  Other Names: Lobeglitazone 0.5mg + Sitagliptin 100mg

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction between lobeglitazone and sitagliptin in healthy male volunteers.

DETAILED DESCRIPTION:
To healthy male subjects of twenty(20), following treatments are administered dosing in each period and wash-out period is a minimum of 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male whose age is over 19 years old when visiting for initial screening test
2. Body mass index(BMI) between 17.5~30.5 kg/m^2 and the body weight must be over 55kg (Body mass index (BMI) = weight (kg) / height (m)^2)
3. A male with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening after examined through hematology test and blood chemistry analysis, urinary test, the electrocardiogram (ECG), and etc.
5. The participants must be volunteered and sign in an informed consent document proven by Chonbuk National University IRB before joining a study to show that he was given informed the purpose of tests and the special characteristics of drugs.
6. The participants must have an ability and willingness to participate throughout the entire trials

Exclusion Criteria:

1. A person who had a history or symptoms of clinically aware of blood, kidney, internal secretion, gastrointestinal, urinary system, cardiovascular, liver, mental, nercous, or allergic(except subclinical seasonal allergies that is not treated at injecion) desease.
2. Who had a gistory of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy)
3. Who had following results after examination

   a. ALT or AST > twice higher than normal value
4. Who constantly intake 210 g/week of alcohol within 6 months of the screening. (a cup of beer (5%) (250 mL) = 10 g, a shot of soju (20%) (50mL) = 8 g, a glass of wine (!2%) (125 mL) = 12g)
5. Who participated other clinical test or took testing bioequivalence drugs in 3 months before the first clinical drug trial.
6. Whose blood pressure ≤ 100 or ≥150(systolic blood pressure) or < 60 or ≥ 100(diastolic blood pressure)
7. Who had a medical history of alcohol and drug abuses.
8. Who had taken a drug that has a control of metabolic rate (activatioh or inhibithion) in 30 days before the first taking of clinical testing durg.
9. WHo smokes more than 20 eigarettes per day.
10. Who took prescribed drugs or over-the-conuter durgs in 10 days before taking of very first clinical testing drug.
11. Who participated in whole blood donation in 2 months before the first taking of clinical testing drugs or platelet donations in 1 month before the first taking to clinical testing drugs.
12. Who has a potent to increase a danger by participating in the clinical trials or sho can interrupt interpretin test results by having serious or chronic medical and mental status or having issues in results of the screening examination.
13. Who has a histroy of an extreme sensitivity of drugs that contain Rosiglitazone or dugs that have similar effect a Rosiglitazone(Pioglitazone), or drugs that contain the ingredients of Sitagliptin or thiazolidinediones drugs.
14. Who has a serious heart failure or a congestive heart failure that must be drug-treated
15. A patient with hepatopathy.
16. A patient with wevere nephropathy.
17. Who has diabetic ketoacidosis or a diaetic coma, or type 1 diabetes, or has history of acute metablic acidosis or ketoacidosis.
18. A patient with serious infectious disease or severe injuries before and after a surgery.
19. Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders.
20. Test subjects who is not willing or unable to comply with guidelines described in this protocol.
21. A person who is not determined unsuitable to participate in this test by the researchers.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUCτ of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
Css,max of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h

SECONDARY OUTCOMES:
Css,min of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
Css,av of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
Tss,max of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
t1/2 of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
CLss/F of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
Vdss/F of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
fluctuation[(Css,max-Css,min)/Css,av] of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h
swing[(Css,max-Css,min)/Css,min] of Lobeglitazone | 1Day 0h, 3Day 0h, 4Day 0h, 5Day 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD,PhD, Study Director — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon SJ, Yu KS, Kim MG. An Assessment of Pharmacokinetic Interaction Between Lobeglitazone and Sitagliptin After Multiple Oral Administrations in Healthy Men. Clin Ther. 2020 Jun;42(6):1047-1057. doi: 10.1016/j.clinthera.2020.04.005. Epub 2020 Apr 30. PMID 32362346